CLINICAL TRIAL: NCT03287544
Title: Effect of a Combined Language Therapy (Linguistic/Communication) on Aphasia After Stroke in Acute Phase: A Prospective, Controlled, Monocentric Pilot Study
Brief Title: Efficacy of a Combined Linguistic/Communication Therapy in Acute Aphasia After Stroke
Acronym: ORACLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC31/16/0018; 2017-A02163-50 (Other: ID-RCB)
Record Dates: First submitted 2017-08-21; First posted 2017-09-19 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Aphasia, Acquired
Keywords: Aphasia; Rehabilitation; Communication; Linguistics
MeSH Terms: conditions — Aphasia; Communication

STUDY DESIGN:
Intervention Model Description: There are two arms in the protocol: one experimental arm corresponding to the "combined" rehabilitation (linguistic/communication) compared with another arm corresponding to the "linguistic" rehabilitation.
  All included patients, after allocation based on aphasia severity to the " combined " and " linguistic " groups, will have a first evaluation (E1: language, neurologic and neuropsychological exams) within 7 days after the onset. Then after a 3 months rehabilitation period they will be assessed (E2: language, neurologic and neuropsychological exams). At 6 months after the onset they will finally have the last assessment (E3: language, neurologic and neuropsychological exams).
Who Masked: Outcomes Assessor
Masking Description: After the allocation in the groups, rehabilitation is not done blindly since the speech therapist knows what activities he offers to patients. However, the evaluations carried out by a speech therapist, are done without the knowledge of the rehabilitation group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined rehabilitation (Experimental): Linguistic training as well as communication training.
  Interventions: Other: Combined rehabilitation
- Linguistic rehabilitation (Active Comparator): Rehabilitation only focused on linguistic processes.
  Interventions: Other: Linguistic rehabilitation

INTERVENTIONS:
Other: Combined rehabilitation — Linguistic training as well as communication training.
  Arms: Combined rehabilitation
Other: Linguistic rehabilitation — Rehabilitation only focused on linguistic processes.
  Arms: Linguistic rehabilitation

SUMMARY:
Linguistic training is traditionally the gold standard for rehabilitation of aphasia after stroke and efficacy criteria count early stage, intensity as well as personalized treatment. To date, no clear evidence showed a specific effect of any therapy in the acute phase of aphasia after stroke. This study aims to compare the effect of a combined therapy (linguistic/communication) versus a linguistic therapy on communication performance in patients in the acute phase of aphasia after a first stroke.

DETAILED DESCRIPTION:
Twenty to 25% of strokes cause aphasia. Speech and language therapy is the well-known standard treatment of aphasia after stroke although it is based on weak scientific evidence. To date, the efficacy criteria of aphasia rehabilitation are early stage, intensity as well as personalized treatment. Usually these patients receive in acute phase a linguistic training focused on the linguistic impairment. This approach is based on the cerebral plasticity postulate. However the superiority of this practice compared to other methods has never been shown. Moreover the benefit of the combination gathering linguistic treatment with communication treatment has to our knowledge never been studied.

In the present study investigators propose to compare the effect of a combined linguistic/communication rehabilitation versus a linguistic treatment. To do so, investigators will recruit patients with aphasia after a first stroke, in the acute phase. After a allocation to the " combined " and " linguistic " groups, all the patients will have a comprehensive language and neuropsychological assessment before and after 3 months of rehabilitation, and finally 6 months after the onset.

The "linguistic" group will have a rehabilitation only focused on linguistic processes whereas the "combined" group will have a linguistic training as well as communication training. The therapy will be personalized and the therapists will exclusively use standardized linguistic and/or communication toolboxes of rehabilitation containing dedicated activities.

ELIGIBILITY:
Inclusion Criteria:

* First stroke
* Inclusion at the acute phase (< 7 days)
* Patient registered at the social security system
* French as usual language
* Aphasia severity score measured by the Boston Diagnostic Aphasia Examination (BDAE) scale ≥ 1 and ≤ 4
* Consent signed by the patient or if not, by the caregiver

Exclusion Criteria:

* Cognitive impairment before the onset (IQCode > 3.4)
* Alcohol or drug addiction
* Untreated psychiatric disease,
* Uncorrected sensory impairment
* Evolutive pathology
* Adults protected by Law
* Participation to another research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Assessment of the communication performance. | Month 3
  Assessed by the Lillois communication test

SECONDARY OUTCOMES:
Assessment of the communication performance. | Month 6
  Assessed by the Lillois communication test
Assessment of the linguistic performance. | Month 3; Month 6
  Assessed by the "Score at understanding task".
Assessment of the quality of life. | Month 3; Month 6
  Assessed by the "Score at a specific quality of life scale ".

CONTACTS AND LOCATIONS:
Overall Officials: Lola Danet, Phd, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hôpital Pierre Paul Riquet, Toulouse, Midi-Pyrénées, France

REFERENCES:
- [Background] Galletta EE, Barrett AM. Impairment and Functional Interventions for Aphasia: Having it All. Curr Phys Med Rehabil Rep. 2014 Jun 1;2(2):114-120. doi: 10.1007/s40141-014-0050-5. PMID 25133085
- [Background] Bhogal SK, Teasell R, Speechley M. Intensity of aphasia therapy, impact on recovery. Stroke. 2003 Apr;34(4):987-93. doi: 10.1161/01.STR.0000062343.64383.D0. Epub 2003 Mar 20. PMID 12649521
- [Background] Tippett DC, Niparko JK, Hillis AE. Aphasia: Current Concepts in Theory and Practice. J Neurol Transl Neurosci. 2014 Jan;2(1):1042. PMID 24904925
- [Background] Jorm AF, Jacomb PA. The Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE): socio-demographic correlates, reliability, validity and some norms. Psychol Med. 1989 Nov;19(4):1015-22. doi: 10.1017/s0033291700005742. PMID 2594878
- [Background] Behrmann M, Lieberthal T. Category-specific treatment of a lexical-semantic deficit: a single case study of global aphasia. Br J Disord Commun. 1989 Dec;24(3):281-99. doi: 10.3109/13682828909019892. PMID 2627547
- [Background] Crosson B. An intention manipulation to change lateralization of word production in nonfluent aphasia: current status. Semin Speech Lang. 2008 Aug;29(3):188-200; quiz C-4. doi: 10.1055/s-0028-1082883. PMID 18720316
- [Background] Jones EV. Building the foundations for sentence production in a non-fluent aphasic. Br J Disord Commun. 1986 Apr;21(1):63-82. doi: 10.3109/13682828609018544. No abstract available. PMID 3730272